CLINICAL TRIAL: NCT05329168
Title: An Open-Label, Multiple-Ascending Dose, Multicenter Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LSVT-1701 as an Add-on to Standard of Care Antibiotics for the Treatment of Complicated Methicillin-Sensitive and -Resistant Staphylococcus Aureus Bacteremia Including Left- and Right-sided Infective Endocarditis
Brief Title: ERAdicate S. Aureus in Patients With Bacteremia and Endocarditis
Acronym: ERASE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: business decision before FPFV; not related to any safety concerns
Sponsor: Lysovant (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSVT-1701-2001
Record Dates: First submitted 2022-03-23; First posted 2022-04-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Bacteremia Due to Staphylococcus Aureus; Left Sided Infective Endocarditis (Disorder); Right Sided Infective Endocarditis (Disorder); Endocarditis Infective
Keywords: Staphylococcus aureus bacteremia; left-sided endocarditis; right-sided endocarditis; SAB
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Intervention Model Description: Sequential ascending-dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential ascending-dose cohort (Experimental): Sequential ascending-dose cohort
  Interventions: Drug: Tonabacase (LSVT-1701)

INTERVENTIONS:
Drug: Tonabacase (LSVT-1701) — 4.5 or 6.0 mg/kg IV once daily for 4 days

SUMMARY:
This study evaluates safety and tolerability of endolysin-derived LSVT-1701 (tonabacase) as an add-on to standard of care (SOC) antibiotic therapy for the treatment of patients with complicated Staphylococcus aureus bacteremia (SAB), including left- and right-sided infective endocarditis (IE).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 90 years
* Index blood culture collection within 96 hours prior to enrollment positive for S. aureus
* Experienced at least one sign or symptom related to SAB within past 96 hours prior to enrollment
* Known or suspected left- and/or right-sided endocarditis by modified Duke criteria and/or known or suspected complicated SAB
* Required duration of SOC antibiotic therapy ≤ 42 days

Exclusion Criteria:

* Previous receipt of LSVT-1701 or CF-301 (exebacase)
* Known hypersensitivity to kanamycin or other aminoglycosides
* Treatment with any potentially effective (anti-S. aureus) systemic antibiotic for > 96 hours within 7 days before enrollment. Exception: Persistent S. aureus bacteremia after 96 hours of prior appropriate systemic antistaphylococcal antibiotic, and/or resistance to the prior systemic antibiotic
* Treatment with dalbavancin or oritavancin within the previous 90 days
* Known or suspected brain abscess or meningitis
* Community acquired pneumonia, nosocomial pneumonia because of pathogens other than S. aureus, or known polymicrobial bacteremia
* Presence of an intravascular infection source or extravascular material that cannot be removed within 96 hours after enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-08-17 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events coded per the Medical Dictionary of Regulatory Activities (MedDRA) v.24.0 [norm] | Up to Day 90±14
Incidence of Grade 3 or Grade 4 toxicity according to modified DAIDS criteria version 2.1 | Up to 14±4 days after end of SOC antibiotic therapy (up to Day 42)
Changes in 12-lead electrocardiogram (ECG) | Day 1 and Day 2

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of LSVT-1701 | Day 4
Area under the concentration-time curve (AUC) of LSVT-1701 | Day 4
Overall clinical response | Day 7, Day 14, after end of SOC antibiotic therapy (up to Day 42), and at test of cure (TOC; 14 days after the EOT)
  Overall clinical response is defined as survival, resolution or improvement of attributable signs and symptoms, no new attributable signs and symptoms, no new foci of S. aureus infection, no change in antibiotics due to non-response, and no further surgery or medical intervention to treat S. aureus.
Microbiological response rate | Days 3, 5, 7, 14, and up to Day 90

OTHER OUTCOMES:
Overall clinical response in patients with left-sided endocarditis | Up to Day 14
  Overall clinical response is defined as survival, resolution or improvement of attributable signs and symptoms, no new attributable signs and symptoms, no new foci of S. aureus infection, no change in antibiotics due to non-response, and no further surgery or medical intervention to treat S. aureus.
Overall clinical response in patients with right-sided endocarditis | Up to Day 14
  Overall clinical response is defined as survival, resolution or improvement of attributable signs and symptoms, no new attributable signs and symptoms, no new foci of S. aureus infection, no change in antibiotics due to non-response, and no further surgery or medical intervention to treat S. aureus.
All-cause mortality | Day 14 and Day 28
Mortality attributable to SAB | Day 14 and Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Lsvt-1701-2001, Butte, Montana, United States

IPD SHARING:
Plan to Share IPD: No